CLINICAL TRIAL: NCT03189524
Title: A Phase I Clinical Study to Investigate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of BTK Inhibitor BGB-3111 in Chinese Patients With B-cell Lymphoma
Brief Title: A Study to Investigate Zanubrutinib in Chinese Participants With B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-1002; CTR20160204 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Results first posted 2021-10-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2021-09

CONDITIONS: B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — zanubrutinib

ARMS (3):
- Part I: 160 mg BID (Experimental): Safety Evaluation: Two regimens of zanubrutinib 320 milligrams (mg) daily (160 mg twice daily [BID]) administered in the morning and at night, or 320 mg (once daily [QD]), and a "3+3" design was adopted for Part I of the study to determine recommended Phase 2 dose (RP2D).
  Interventions: Drug: Zanubrutinib
- Part I: 320 mg QD (Experimental): Safety Evaluation: Two regimens of zanubrutinib 320 mg daily (160 mg BID, administered in the morning and at night, or 320 mg QD) and a "3+3" design was adopted for Part I of the study to determine RP2D.
  Interventions: Drug: Zanubrutinib
- Part II: 160 mg BID (Experimental): Dose Expansion: The RP2D determined in Part I was used in Part II to further evaluate the preliminary anti-tumor effects of zanubrutinib in Chinese participants with follicular lymphoma (FL) or marginal zone lymphoma (MZL).
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib is a white to off-white solid that is slightly hygroscopic. The drug product was formulated as 20-mg (blue, size 3) and 80-mg (white, size 0) hard gelatin, opaque oral capsules. Zanubrutinib is classified as a Biopharmaceutics Classification System Class II compound.
  Other Names: BGB-3111

SUMMARY:
This phase I clinical study was to investigate the safety, tolerability, and pharmacokinetics/pharmacodynamics of Bruton tyrosine kinase (BTK) inhibitor zanubrutinib (BGB-3111) in Chinese participants with B-cell lymphoma by conducting in two stages, the first stage being the safety assessment of dose and the second stage being the dose expansion.

Part I: Safety evaluation - according to the results of preclinical toxicological trials and the results of the phase I clinical study conducted in Australia and New Zealand, two regimens of zanubrutinib 320 milligrams (mg) daily (160 mg twice daily [BID]), administered in the morning and at night, or 320 mg once daily [QD]) and "3+3" design was adopted for the assessment. The recommended dose and method of administration of the phase II clinical study was determined according to the Part I results.

Part II: Dose expansion - this stage was to further evaluate the preliminary anti-tumor effects of zanubrutinib in Chinese participants with follicular lymphoma (FL) or marginal zone lymphoma (MZL), approximately 20 participants with relapsed or refractory FL or MZL were to be enrolled. The recommended Phase 2 dose (RP2D) was used in Part II.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and women between the age of 18-75 years.
* Participants with B-cell lymphoma (defined by World Health Organization classification) refractory or relapsed following at least one line of therapy.
* Judged by the investigator as requiring treatment.
* Eastern Cooperative Oncology Group performance status of 0-1.
* Life expectancy of at least 4 months.
* Adequate hematological function.
* Adequate renal function.
* Adequate liver function.
* Adequate coagulation function.
* Female participants of childbearing potential and non-sterile males must have practiced at least one of the following methods of birth control with partner(s) throughout the study and for 90 days after discontinuing study drug: total abstinence from sexual intercourse, double-barrier contraception, intrauterine device or hormonal contraceptive initiated at least 3 months prior to first dose of study drug.
* Male participants must not have donated sperm from start of study drug administration, until 90 days after discontinuation of treatment.

Key Exclusion Criteria:

* With central nervous system involvement of the disease.
* The pathological type of the disease had disease transformation.
* Had underdone allogeneic hematopoietic stem cell transplantation.
* Had received corticosteroid anti-neoplastic treatment within 7 days before the first dose, has received radiotherapy and chemotherapy within 4 weeks before the first dose or has received treatment with monoclonal antibody within 4 weeks before the first dose.
* Had received BTK inhibitor treatment prior to enrollment.
* Had received chemotherapy and has not yet recovered from toxicity
* Had received Chinese herbal medicine as anti-neoplastic therapy within 4 weeks before starting study treatment.
* History of other malignancies within 2 years before study.
* With uncontrolled systemic infection.
* Major surgery in the past 4 weeks.
* With known HIV, or active hepatitis B or hepatitis C virus infection.
* With cardiovascular disease of New York Heart Association Classification ≥ 3.
* Significant electrocardiogram abnormalities.
* Significant active renal, neurologic, psychiatric, hepatic or endocrinologic disease that in the investigator's opinion would adversely impact on his/her participation in the study.
* Inability to comply with study procedures.
* Was currently taking anticoagulant drugs.
* Was currently taking potent cytochrome P450 3A inhibitor or inducer.
* Had stroke or cerebral hemorrhage within 6 months before enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may have applied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jun Zhu, BS, Jianyong Li, MD, Jianfeng Zhou, Yuqin Song, MD, Junyuan Qi, Wei Xu, Dengju Li, MD, Mingyuan Sun, Ling Xue, PhD, Liudi Yang, Yinwei Zhang, Lai Wang, PhD, Jane Huang, MD, Shibao Feng, PhD, Lugui Qiu, MD. BGB-3111, a Highly Specific BTK Inhibitor, Is Well Tolerated and Highly Active in Chinese Patients with Relapsed/Refractory B-Cell Malignancies: Initial Report of a Phase 1 Trial in China. Blood. 2017; 130(1): 5347. https://doi.org/10.1182/blood.V130.Suppl_1.5347.5347
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Xu W, Yang S, Tam CS, Seymour JF, Zhou K, Opat S, Qiu L, Sun M, Wang T, Trotman J, Pan L, Gao S, Zhou J, Zhou D, Zhu J, Song Y, Hu J, Feng R, Huang H, Su D, Shi M, Li J. Zanubrutinib Monotherapy for Naive and Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: A Pooled Analysis of Three Studies. Adv Ther. 2022 Sep;39(9):4250-4265. doi: 10.1007/s12325-022-02238-7. Epub 2022 Jul 28. PMID 35900694
- [Derived] Song Y, Sun M, Qi J, Xu W, Zhou J, Li D, Li J, Qiu L, Du C, Guo H, Huang J, Tang Z, Ou Y, Wu B, Yu Y, Zhu J. A two-part, single-arm, multicentre, phase I study of zanubrutinib, a selective Bruton tyrosine kinase inhibitor, in Chinese patients with relapsed/refractory B-cell malignancies. Br J Haematol. 2022 Jul;198(1):62-72. doi: 10.1111/bjh.18162. Epub 2022 Apr 5. PMID 35383885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 4 centers in China, all of which enrolled participants. The first participant was dosed on 05 July 2016. As of the final database lock (15 October 2020), 44 participants were enrolled and treated with zanubrutinib (BGB-3111). Once the final analysis was completed, the study was terminated and all participants who were still on treatment were transferred to long term extension study.
Groups:
- Part I: 160 mg BID: Safety Evaluation: The participants in this dose regimen received zanubrutinib 320 milligrams (mg) (160 mg twice daily [BID], administered in the morning and at night) and a "3+3" design was adopted for Part I of the study to determine RP2D.
- Part I: 320 mg QD: Safety Evaluation: The participants in this dose regimen received zanubrutinib 320 mg daily (320 mg once daily [QD]) and a "3+3" design was adopted for Part I of the study to determine RP2D.
Period: Overall Study
Arm/Group | Part I: 160 mg BID | Part I: 320 mg QD | Part II: 160 mg BID
Started | 11 | 10 | 23
Received at Least 1 Dose of Study Drug | 11 | 10 | 23
Completed | 0 | 0 | 0
Not Completed | 11 | 10 | 23
Not completed — Study terminated by Sponsor after final analysis and all remaining participants transferred to LTE | 7 | 5 | 11
Not completed — Death | 2 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 8
Not completed — Withdrawal by Subject | 1 | 1 | 3
Not completed — Progressive Disease | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part I: 160 mg BID: Safety Evaluation: The participants in this dose regimen received zanubrutinib 320 mg daily (160 mg BID, administered in the morning and at night) and a "3+3" design was adopted for Part I of the study to determine RP2D.
- Part I: 320 mg QD: Safety Evaluation: The participants in this dose regimen received zanubrutinib 320 mg daily (320 mg QD) and a "3+3" design was adopted for Part I of the study to determine RP2D.
- Part II: 160 mg BID: Dose Expansion: The RP2D determined in Part I was used in Part II to further evaluate the preliminary anti-tumor effects of zanubrutinib in Chinese participants with FL or MZL.
- Total: Total of all reporting groups
Arm/Group | Part I: 160 mg BID | Part I: 320 mg QD | Part II: 160 mg BID | Total
Number analyzed (Participants) | 11 | 10 | 23 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (10.65) | 52.1 (10.57) | 48.4 (11.85) | 50.1 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 15 | 20
  Male | 9 | 7 | 8 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 10 | 23 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part I: Number Of Participants Experiencing Treatment-emergent Adverse Events And Treatment-emergent Serious Adverse Events
Description: All adverse events were treatment emergent and were defined as an adverse event with a reported onset time or increase in severity after the initial dose of study drug and within 30 days after the last dose of study drug or initiation of new anticancer therapy, whichever was sooner. A serious adverse event was any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is significant medical event requiring intervention. All toxicity and adverse events were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.03 (NCI-CTCAE v4.03) grading criteria. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From the date of informed consent until 30 +/- 7 days after treatment discontinuation (up to 4 years and 1 month)
Population: Safety Analysis Set: Included all participants who received ≥ 1 dose of zanubrutinib. The Safety Analysis Set was used for all summaries (except DLT and PK).
Measure: Count of Participants; unit: Participants
Arm/Group | Part I: 160 mg BID | Part I: 320 mg QD
Number analyzed (Participants) | 11 | 10
Participants
  Participants with ≥ 1 adverse event | 11 | 10
  Participants with serious adverse events | 2 | 2

2. Primary Outcome: Part II: Overall Response Rate (ORR) Of Zanubrutinib In Participants With FL And MZL
Description: Overall response in overall response rate (ORR) was defined as a participant's best overall response: CR or PR for NHL participants; CR, complete remission with incomplete blood count recovery, nodular PR, PR, or PR with lymphocytosis for the CLL participants; CR, very good PR, PR, or minor response for the Waldenström macroglobulinemia participants. ORR was defined as the percentage of participants who achieved an overall response.
Time Frame: Up to 4 years and 1 month
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Percentage of Participants | 30.4 [13.2 to 52.9]

3. Primary Outcome: Part II: Complete Response Rate (CRR) Of Zanubrutinib In Participants With FL And MZL
Description: CRR was defined as the percentage of participants who achieved CR as the best overall response.
Time Frame: Up to 4 years and 1 month
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Percentage of Participants | 13 [2.8 to 33.6]

4. Primary Outcome: Part II: Partial Response Rate (PRR) Of Zanubrutinib In Participants With FL And MZL
Description: PRR was defined as the percentage of participants who achieved PR or higher as the best overall response.
Time Frame: Up to 4 years and 1 month
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Percentage of Participants | 30.4 [13.2 to 52.9]

5. Primary Outcome: Part II: Duration of Response (DOR) Of Zanubrutinib In Participants With FL And MZL
Description: Duration of response for responders (those who achieved an overall response of PR or better) was defined as the time interval (in number of days) between the date of the earliest qualifying response and the date of progressive disease or death for any cause (whichever occurs earlier). Duration of response analysis included only responders.
Time Frame: Up to 4 years and 1 month
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Months | 11.2 [2.8 to NA] — NA = Not Estimable due to insufficient number of participants with events

6. Primary Outcome: Part II: Progression Free Survival (PFS) Of Zanubrutinib In Participants With FL And MZL
Description: Progression-free survival was defined as the time (in months) from the date of first study treatment to disease progression or death (due to any cause), whichever occurred first. For purposes of calculating PFS, the start date of progressive disease was the date at which progression was first observed. The duration and primary analysis of PFS was right-censored for participants who met 1 of the following conditions: 1) no baseline disease assessments; 2) starting a new anticancer therapy before documentation of disease progression or death; 3) death or disease progression immediately after more than 1 consecutively missed disease assessment visit; and 4) alive without documentation of disease progression before the data cutoff date.
Time Frame: Up to 4 years and 1 month
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Months | 5.5 [4.6 to 16.4]

7. Secondary Outcome: Part I and Part II: Area Under The Plasma Concentration-time Curve From Zero To The Last Measurable Concentration (AUClast) For Single-dose Zanubrutinib
Time Frame: Part 1 and 2 : Week 1 day1 Pre-dose, 0.5, 1, 2, 3, 4, 6 (part2 only), 8, 12 and 24 hours, and Week 2-day 1 Pre-dose, 0.5, 1, 2, 3, 4, 6 (part2 only), 8, and 12 hours (part2 only), and Week 5 and Week 9 Day 1 Pre-dose
Population: The PK analysis set included all participants who received ≥ 1 dose of zanubrutinib. The analysis was pre-specified to be a pooled analysis by dose level; therefore, data by individual arms was not analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter*hour
Groups:
- 160 mg BID: Part I: Zanubrutinib 320 mg daily (160 mg BID, administered in the morning and at night) and a "3+3" design was adopted for Part I of the study to determine RP2D.
  Part II: The RP2D determined in Part I was used in Part II to further evaluate the preliminary anti-tumor effects of zanubrutinib in Chinese participants with FL or MZL.
- 320 mg QD: Part I: Zanubrutinib 320 mg daily (QD) and a "3+3" design was adopted for Part I of the study to determine RP2D.
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 34 | 10
nanogram/milliliter*hour | 981.6 (619.6) | 1404 (560.7)

8. Secondary Outcome: Part I and Part II: Area Under The Plasma Concentration-time Curve Zero To Infinity (AUC0-inf) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram/milliliter*hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 32 | 9
nanogram/milliliter*hour | 1025 (633.5) | 1537 (519.0)

9. Secondary Outcome: Part I And Part II: Maximum Plasma Concentration (Cmax) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 34 | 10
nanogram/milliliter | 319 (217) | 409 (149)

10. Secondary Outcome: Part I and Part II: Time To Maximum Plasma Concentration (Tmax) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 34 | 10
hour | 2.00 [0.42 to 5.98] | 2.50 [1.00 to 4.00]

11. Secondary Outcome: Part I and Part II: Apparent Terminal Half Life (t1/2) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 32 | 9
hour | 2.27 (1.21) | 3.43 (2.23)

12. Secondary Outcome: Part I and Part II: Apparent Plasma Clearance (CL/F) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: The PK analysis set included all participants who received ≥ 1 dose of zanubrutinib. The analysis was pre-specified to be a pooled analysis by dose level; therefore, data by individual arms was not analyzed. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 32 | 9
liter/hour | 251 (194) | 235 (93.7)

13. Secondary Outcome: Part I and Part II: Terminal Apparent Volume Of Distribution (Vz/F) For Single-dose Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: liter
Groups:
- 160 mg: Part I: Zanubrutinib 320 mg daily (160 mg BID, administered in the morning and at night) and a "3+3" design was adopted for Part I of the study to determine RP2D.
  Part II: The RP2D determined in Part I was used in Part II to further evaluate the preliminary anti-tumor effects of zanubrutinib in Chinese participants with FL or MZL.
Arm/Group | 160 mg | 320 mg QD
Number analyzed (Participants) | 32 | 9
liter | 713 (512) | 1120 (738)

14. Secondary Outcome: Part I and Part II: Area Under The Plasma Concentration-time Curve For Steady State (AUCss) Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram/milliliter*hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 33 | 8
nanogram/milliliter*hour | 738.3 (425.2) | 1277 (607.4)

15. Secondary Outcome: Part I and Part II: Maximum Plasma Concentration At Steady State (Cmax,ss) For Zanubrutinib
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 33 | 10
nanogram/milliliter | 257 (147) | 389 (185)

16. Secondary Outcome: Part I and Part II: Time To Steady Plasma Concentration (Tmax,ss) For Zanubrutinib
Time Frame: as for outcome 7
Measure: Median (Full Range); unit: hour
Arm/Group | 160 mg BID | 320 mg QD
Number analyzed (Participants) | 33 | 10
hour | 2.00 [0.43 to 2.93] | 2.0 [1.00 to 3.27]

17. Secondary Outcome: Part I: Percentage of BTK Occupied In Peripheral Blood Mononuclear Cells In Participants Who Received Zanubrutinib
Description: The percentage of BTK occupied in peripheral blood mononuclear cells was evaluated as a biomarker for the inhibition of BTK on specified days and the average value is reported.
Time Frame: DLT Period: Days 1 and 2 of Week 1 and Day 1 of Week 2
Population: DLT Evaluable Set: Included all participants who received ≥ 75% of the planned doses of treatment during the DLT observation period (Day 28).Only participants with sufficient sample availability were used in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage
Groups:
- Part I: 160 mg BID or 320 mg QD: Safety Evaluation: The participants in this dose regimen received zanubrutinib 320 mg daily (160 mg BID, administered in the morning and at night) or 320 mg QD and a "3+3" design was adopted for Part I of the study to determine RP2D.
Arm/Group | Part I: 160 mg BID or 320 mg QD
Number analyzed (Participants) | 13
Percentage | 96.69 (5.297)

18. Secondary Outcome: Part II: Number Of Participants Experiencing Treatment-emergent Adverse Events And Treatment-emergent Serious Adverse Events
Description: All adverse events are treatment emergent, defined as an adverse event with a reported onset time or increase in severity after the initial dose of study drug and within 30 days after the last dose of study drug or initiation of new anticancer therapy, whichever was sooner. A serious adverse event was any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is significant medical event requiring intervention. All toxicity and adverse events were assessed according to the NCI-CTCAE v4.03 grading criteria. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From the date of informed consent until 30 +/- 7 days after treatment discontinuation (up to 4 years and 1 month)
Measure: Count of Participants; unit: Participants
Arm/Group | Part II: 160 mg BID
Number analyzed (Participants) | 23
Participants
  Participants with ≥ 1 adverse event | 22
  Participants with serious adverse events | 5

ADVERSE EVENTS:
Time Frame: From the date of informed consent until 30 +/- 7 days after treatment discontinuation (up to 4 years and 1 month)
Arm/Group | Part I: 160 mg BID | Part I: 320 mg QD | Part II: 160 mg BID
All-Cause Mortality (participants affected / at risk) | 2/11 | 3/10 | 1/23
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/10 | 5/23
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: 160 mg BID (N=11) | Part I: 320 mg QD (N=10) | Part II: 160 mg BID (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Pleural infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cholesterin granuloma of middle ear (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I: 160 mg BID (N=11) | Part I: 320 mg QD (N=10) | Part II: 160 mg BID (N=23)
Neutrophil count decreased (Investigations) | 8 | 7 | 9
White blood cell count decreased (Investigations) | 3 | 3 | 9
Platelet count decreased (Investigations) | 4 | 2 | 4
Weight increased (Investigations) | 2 | 3 | 3
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 2
Weight decreased (Investigations) | 0 | 1 | 3
White blood cells urine positive (Investigations) | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 1 | 0
Blood urine present (Investigations) | 0 | 1 | 2
White blood cell count increased (Investigations) | 0 | 1 | 2
Blood fibrinogen decreased (Investigations) | 2 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 5 | 5
Pneumonia (Infections and infestations) | 3 | 3 | 3
Nasopharyngitis (Infections and infestations) | 5 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 2 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 8
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 2
Platelet dysfunction (Blood and lymphatic system disorders) | 3 | 1 | 2
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Purpura (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 4 | 3 | 2
Haemoglobinuria (Renal and urinary disorders) | 2 | 1 | 3
Proteinuria (Renal and urinary disorders) | 2 | 1 | 2
Leukocyturia (Renal and urinary disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 3 | 1
Asthenia (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03189524/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03189524/SAP_001.pdf